CLINICAL TRIAL: NCT03872050
Title: Deep Phenotyping of Rosacea and Migraine
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Nita Katarina Frifelt Wienholtz, Principal Investigator, Medical Doctor, PhD Fellow, Danish Headache Center
Other Study IDs: RosMigInterview
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Migraine; Rosacea
MeSH Terms: conditions — Migraine Disorders; Rosacea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Mouthswab for DNA-sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rosacea: Patients who have been diagnosed with rosacea
  Interventions: Diagnostic Test: No intervention apart from tests, including interview
- Migraine: Patients who have been diagnosed with migraine
  Interventions: Diagnostic Test: No intervention apart from tests, including interview

INTERVENTIONS:
Diagnostic Test: No intervention apart from tests, including interview — No interventions

SUMMARY:
This study aims to deep phenotype patients with rosacea and migraine

DETAILED DESCRIPTION:
Rosacea and migraine are common disorders that overlap in epidemiology, symptoms, trigger factors, and distribution in the trigeminal area. Recent studies establish a connection between the two disorders, which needs to be investigated.

The purpose of this study is investigate the link between the two disorders by deep phenotyping through semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis with either rosacea and/or migraine

Exclusion Criteria:

* does not want to participate
* cannot co-operate to investigation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rosacea
  * patients invited to participate through 3 different clinics in Copenhagen and Zealand, Denmark
  Migraine
  * patients attending the outpatient clinic of the Danish Headache Center invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of migraine in rosacea cohort | 60 minutes
  Prevalence of patients in rosacea cohort who fulfill diagnostic criteria for migraine
Prevalence of rosacea in migraine cohort Prevalence of rosacea in migraine cohort | 60 minutes
  Prevalence of patients in migraine cohort who fulfill diagnostic criteria for rosacea

SECONDARY OUTCOMES:
Prevalence of migraine subtypes in rosacea cohort | 60 minutes
  Prevalence of patients in rosacea cohort who fulfill diagnostic criteria for subtypes of migraine according to international headache society classification
Prevalence of rosacea subtypes in migraine cohort | 60 minutes
  Prevalence of patients in migraine cohort who fulfill diagnostic criteria for subtypes of rosacea

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, PhD, DMSc, Principal Investigator — Professor
Locations (1):
- Danish Headache Center, Glostrup, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wienholtz NKF, Christensen CE, Ashina H, Jorgensen NR, Egeberg A, Thyssen JP, Ashina M. Elevated plasma levels of calcitonin gene-related peptide in individuals with rosacea: A cross-sectional case-control study. J Eur Acad Dermatol Venereol. 2025 Jan;39(1):181-188. doi: 10.1111/jdv.19954. Epub 2024 Apr 1. PMID 38558478
- [Derived] Wienholtz NKF, Christensen CE, Haugaard JH, Zhang DG, Ashina M, Thyssen JP, Egeberg A. Cohort profile: COpenhagen ROsacea COhort (COROCO) and COpenhagen MIgraine COhort (COMICO). BMJ Open. 2020 Aug 20;10(8):e039445. doi: 10.1136/bmjopen-2020-039445. PMID 32819957